CLINICAL TRIAL: NCT06895499
Title: A Phase I/II, Open-Label, Dose-Escalation Clinical Trial to Evaluate the Safety and Efficacy of HB0043 (Bispecific Antibody Targeting IL-17A and IL-36R) in Adult Patients With Moderate to Severe Hidradenitis Suppurativa (HS).
Brief Title: Efficacy, Safety, and Tolerability of HB0043 in Hidradenitis Suppurativa Patients.
Acronym: HB0043-HS-0-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Dermatology Hospital affiliated to Shandong First Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HB0043-HS-0-01
Record Dates: First submitted 2025-03-07; First posted 2025-03-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HB0043: Low dose (Experimental): Participants assigned to arm 1 will receive a low dose of HB0043 via intravenous infusion every two weeks starting from week 0. The dose of HB0043 will adjusted to high dose at weeks 10, and the frequency remains Q2W. The frequency will adjusted to Q4W from weeks16, the last administration is weeks 20.
  Interventions: Drug: HB0043
- HB0043: Medium dose (Experimental): Participants assigned to Arm 2 will receive a medium dose of HB0043 via intravenous infusion every two weeks, commencing at week 0, and then at weeks 16 and 20.
  Interventions: Drug: HB0043
- HB0043: High dose (Experimental): Participants assigned to Arm 3 will receive a high dose of HB0043 via intravenous infusion every two weeks, commencing at week 0, and then at weeks 16 and 20.
  Interventions: Drug: HB0043

INTERVENTIONS:
Drug: HB0043 — Low dose
  Arms: HB0043: Low dose
Drug: HB0043 — Medium dose
  Arms: HB0043: Medium dose
Drug: HB0043 — High dose
  Arms: HB0043: High dose

SUMMARY:
The purpose of this study is to assess efficacy safety and tolerability of HB0043 in adult patients with moderate to severe HS.

DETAILED DESCRIPTION:
The total duration of the study is 28 weeks and consists of: Screening (up to 4 weeks), Treatment Period (20 weeks) and Safety Follow-Up (treatment-free follow-up for 4 weeks).

Participants who prematurely discontinue study treatment are encouraged to remain in the study. Participants who do not wish to remain in the study will enter a 4-week Safety Follow-Up period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understand the research procedure of this study and provide written informed consent; 2. Male or female, age 18 years or greater; 3. Diagnosis of HS with a disease duration of at least 6 months before screening; 4. Moderate to severe HS, concurrently meeting the following three criteria:

  1. HS lesions in at least 2 distinct anatomic area;
  2. One of the HS lesions must be Hurley Stage II or Hurley Stage III;
  3. Total abscess and inflammatory nodule (AN) count of greater than or equal to 3; 5. Acceptance by the patient, of childbearing age, to use safe contraceptive methods throughout the study, including six months of follow-up.

Exclusion Criteria:

* 1. Participants with known hypersensitivity to HB0043 or any of its excipients; 2. Participant has a draining fistula count of ≥20 at the Screening Visit; 3. Presence of other active autoimmune diseases except HS, including but not limited to psoriasis, psoriatic arthritis, rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, and uveitis; 4. Participant has any other active skin disease or condition that may interfere with the assessment of hidradenitis suppurativa; 5. History of lymphoproliferative disorders or any known malignancy within five years prior to the Screening Visit (excluding treated and cured cutaneous squamous cell carcinoma, basal cell carcinoma, carcinoma uterine in situ, or intraductal breast cancer in situ); 6. History of recurrent or recent serious infection; 7. Participant has active tuberculosis (TB) or concurrent treatment for latent TB or evidence of hepatitis B virus (HBV) or hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection; 8. Pregnant or lactating women; 9. Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of HB0043 in Patients with Moderate to Severe HS | From randomization to end of study, assessed up to 24 weeks.
  The incidence rate, characteristics, relevance, and severity of treatment-emergent adverse events (TEAEs) experienced by subjects during the treatment period.

SECONDARY OUTCOMES:
Percentage of participants achieving HiSCR | Week 16 and 24
  Percentage of participants achieving HiSCR at Week 12 was reported. For this score participants were defined as achievers or non-achievers. The positive HiSCR score was defined as a greater than or equal to (>=) 50% reduction in inflammatory lesion AN count (sum of abscesses and inflammatory nodules), and no increase in abscesses or draining fistulas in hidradenitis suppurativa compared with the lesions counted on visit 1 (baseline).
Change From Baseline in Inflammatory Lesion (Abscesses and Inflammatory Nodules) Count | Week 16 and 24
  The sum of abscesses and inflammatory nodules was measured for each participant to assess change in inflammatory lesion counts.
Change From Baseline in the number of lesions | Week 16 and 24
  The number of lesions refers to the total sum of abscesses, iInflammatory nodules, and draining fistulas count.
Percentage of Participants Achieving ≥ 30% Reduction and ≥ 1 Unit Reduction From Baseline in PGA-NRS | Week 16 and 24
  PGA-NRS is evaluated based on worst skin pain in a 24-hour recall period (maximal daily pain), ranging from 0 (no skin pain) to 10 (skin pain as bad as you can imagine). The percentage of participants who achieved at least 30% reduction and at least 1 unit reduction from Baseline in the PGA-NRS.
Percentage of participants achieving HiSCR75 | Week 16 and 24
  HiSCR75 is defined as at least a 75% reduction from Baseline in the total abscess and inflammatory nodule [AN] count, with no increase from Baseline in abscess or draining tunnel count
Change in absolute score from Baseline in International Hidradenitis Suppurativa Severity Score System (IHS4) | Week 16 and 24
  Change from baseline in IHS4. IHS4 score is calculated by the number of nodules (multiplied by 1) + the number of abscesses (multiplied by 2) + the number of draining tunnels (multiplied by 4).
  A total score of 3 or less signifies mild, 4-10 signifies moderate and 11 or higher signifies severe disease.
Serum HB0043 concentrations throughout the study | From randomization to end of study, assessed up to 24 weeks.
Incidence of anti-HB0043 antibody positive response throughout the study | From randomization to end of study, assessed up to 24 weeks.
Percentage of participants achieving HiSCR90 | Week 16 and 24
  HiSCR90 is defined as at least a 90% reduction from Baseline in the total abscess and inflammatory nodule [AN] count, with no increase from Baseline in abscess or draining tunnel count
Percentage of participants achieving HiSCR100 | Week 16 and 24
  HiSCR100 is defined as at least a 100% reduction from Baseline in the total abscess and inflammatory nodule [AN] count, with no increase from Baseline in abscess or draining tunnel count
Change of the most severe Patient's Global Assessment of Skin Pain (PGA Skin Pain) within the past 24 hours | Week 16 and 24
  The change from baseline in the most severe PGA Skin Pain (NRS score) within the past 24 hours
Dermatology Life Quality Index (DLQI) | Week 16 and 24
  Percentage of participants achieving a DLQI total reduction of ≥4 minimal clinically important difference among participants with a baseline DLQI ≥4. DLQI produces a numeric score that can range from 0 to 30. A higher score indicates greater health related quality of life impairment.
hange of Hidradenitis Suppurativa Area and Severity Index Revised (HASI-R) | Week 16 and 24
  Change from baseline in HASI-R
Change of HIDRA score | Week 16 and 24
  Change from baseline in HIDRA score
Long-term efficacy of sonelokimab: Hidradenitis Suppurativa Quality of Life (HiSQOL) | Week 16 and 24
  Change from baseline in HiSQOL total score
Change of Numerical Rating Scale (NRS) | Week 16 and 24
  Percentage of participants achieving a ≥3-unit reduction from baseline in the NRS
Pharmacodynamic indicators include but are not limited to IL-17 and IL-36. | From randomization to end of study, assessed up to 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Hospital affiliated to Shandong First Medical University, Jinan, Shandong, China